CLINICAL TRIAL: NCT00001573
Title: A Phase I Study of SU101 in Pediatric Patients With Refractory Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970087; 97-C-0087
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Glioma; Sarcoma
Keywords: Glioma; PDGF; Pharmacokinetics; Sarcoma; Toxicity
MeSH Terms: conditions — Glioma; Sarcoma | interventions — Leflunomide

INTERVENTIONS:
Drug: SU101

SUMMARY:
A dose escalation scale consisting of 5 dosage levels is being used to determine the maximum tolerated dose (MTD) of SU101. A minimum of 3 and a maximum of 6 patients will be enrolled at each dose level. MTD is defined as the dose level immediately below that at which 2 or more patients exhibit dose limiting toxicity.

Each treatment cycle is 21 days. Patients receive a 96 hour continuous IV infusion of SU101 on days 1-4.

DETAILED DESCRIPTION:
SU101 is a member of a novel class of antineoplastic agents, platelet-derived growth factor (PDGF) receptor inhibitors. Preclinical data suggests that SU101 might be an effective agent against neuroglial tumors as well as a variety of sarcomas. A pediatric phase I trial of SU101 in children with these malignancies will be conducted to find the maximum tolerated dose of SU101 and define the toxicity profile of this agent. In addition, we will define the pharmacokinetics of SU101 and its active metabolite SU0020 in pediatric patients and gather preliminary information regarding response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven primary CNS malignancy, neuroblastoma or sarcoma that is refractory to standard therapy or for which no standard therapy exists and disease can not be cured by surgery.

PRIOR/CONCURRENT THERAPY:

Recovered from toxic affects of all prior therapy.

No investigational agent within past 2 weeks.

BIOLOGY THERAPY: Not specified.

CHEMOTHERAPY:

No myelosuppressive therapy within past 3 weeks.

No nitrosourea within past 6 weeks.

ENDOCRINE THERAPY: If receiving dexamethasone dose must be stable for at least 2 weeks.

RADIOTHERAPY: Not specified.

SURGERY: Not specified.

PATIENT CHARACTERISTICS:

Age: 3 to 21.

Performance status: ECOG 0-2.

Life expectancy: At least 8 weeks.

HEMATOPOIETIC:

AGC greater than 1500/mm(3).

Hemoglobin greater than or equal to 8.0 g/dL percent.

Platelet count greater than 100,000/mm(3).

For patients with bone marrow involvement or history of bone marrow transplantation or craniospinal radiotherapy: AGC greater than 750/mm(3), Hemoglobin greater than 6.0 g/dL, Platelet count greater than 50,000/mm(3).

HEPATIC:

SGOT, SGPT or alkaline phosphatase less than 3 times upper limit of normal.

Bilirubin no less than or equal to 1.5 times upper limit of normal.

RENAL:

Ages 3-5 Creatinine no greater than 0.8 mg/dL.

Ages 5-10 Creatinine no greater than 1.0 mg/dL.

Ages 10-15 Creatinine no greater than 1.2 mg/dL.

Ages 16-21 Creatinine no greater than 1.5 mg/dL.

OTHER:

All patients or their legal guardians (if the patient is under 18 years old) must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study.

For patients with brain tumors who are over 18 years of age, a DPA should be signed.

Not pregnant or nursing.

Not allergic to etoposide.

No acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risks associated with study participation/study drug administration or may interfere with the interpretation of study results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1997-03; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Westermark B, Heldin CH, Nister M. Platelet-derived growth factor in human glioma. Glia. 1995 Nov;15(3):257-63. doi: 10.1002/glia.440150307. PMID 8586462
- [Background] Maxwell M, Naber SP, Wolfe HJ, Galanopoulos T, Hedley-Whyte ET, Black PM, Antoniades HN. Coexpression of platelet-derived growth factor (PDGF) and PDGF-receptor genes by primary human astrocytomas may contribute to their development and maintenance. J Clin Invest. 1990 Jul;86(1):131-40. doi: 10.1172/JCI114675. PMID 2164040
- [Background] Matsui T, Sano K, Tsukamoto T, Ito M, Takaishi T, Nakata H, Nakamura H, Chihara K. Human neuroblastoma cells express alpha and beta platelet-derived growth factor receptors coupling with neurotrophic and chemotactic signaling. J Clin Invest. 1993 Sep;92(3):1153-60. doi: 10.1172/JCI116684. PMID 8376577